CLINICAL TRIAL: NCT03265626
Title: Community Based Intervention to Prevent Domestic Violence Against Women in Ethiopia; a Protocol for Quasi-Experimental Implementation Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Haramaya Unversity (Other)
Collaborators: World Health Organization (Other); University of Ghana (Other)
Responsible Party: Principal Investigator, Agumasie Semahegn, PhD Candidate, Haramaya Unversity
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HaramayaU
Record Dates: First submitted 2017-08-26; First posted 2017-08-29 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Domestic Violence Against Women; Community-based Prevention; Interevntion Implementation

STUDY DESIGN:
Intervention Model Description: Community based three arm quasi-experimental design will be employed using mixed methods (quantitative and qualitative). Study participants will be allocated to the intervention and control groups to piloting the feasibility and effectiveness of community based intervention to avert domestic violence against women (15-49 years). Married or cohabited women, husbands/partner, community representatives (such as leaders/local politicians, religious leaders and elders), health care providers, police, women association and women affair office representatives will be involved in this implementation research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comprehensive (Intervention 1) (Experimental): A total of 586 study particpnats will be invloved on this comprehensive (main) experiment group.This arm will receive a comprehensive intervention package that include advocacy to local governors, community mobilization, awareness creation, training of community representatives and engagement partners. community mobilization through engaging husband as change agent to avert domestic violence in collaboration with community Health Extension Workers. The intervention will target married or cohabited women, partner, and community representatives (religious leaders, and elders). The intervention will be focused on physical, psychological and sexual violence, decision making, negotiation, communication on household matters, gender equality and equity norms, and their relationship with women's health. In addition, massive public information dissemination will be done in the intervention community.
  Interventions: Behavioral: Intervention 1: Comprehensive preventive intervention
- Intervention 2 (Active Comparator): A total of 586 study particpnats will be invloved on this active comprator group. The intervention package such as advocacy to local governors, community mobilization, awareness creation and training of community representatives will be carried out for 12 months period.The main diffrence from the arm-1,here is no husband involvment in the interevntion targets. This intervention will be targeted married and cohabited women and community representatives (religious leaders, health care provider, police, politicians and associations). This group of participant will be selected from one urban and one rural Kebele in Banja District. Same tool and approach will be used to track the intervention progress.
  Interventions: Behavioral: Intervention 2: Awareness creation and community mobilization
- Control/Comparator (Other): A total of 586 study partipants will be assigned to the control group that will receive the existing standard services from both urban and rural kebeles of the Guagussa Shikudad district. As comparator purpose, baseline and endline evaluation data will be taken.
  -No intervention package but standard service will be maintained
  Interventions: Other: available standard care

INTERVENTIONS:
Behavioral: Intervention 1: Comprehensive preventive intervention — aims to implement the existing evidence and policy documents Advocacy workshop to politicians, Community mobilization, Awareness creation on women,training community representative, Husband participation
  Arms: Comprehensive (Intervention 1)
Behavioral: Intervention 2: Awareness creation and community mobilization — Advocacy politicians, Community mobilization, Awareness creation to women, Training community representative
  Arms: Intervention 2
Other: available standard care — The standard care will be maintained but no other additional intevvenion designed by this study
  Arms: Control/Comparator

SUMMARY:
Violence against women is a well understood devastating global pandemic, and human right violation. One in three women experienced intimate partner violence worldwide. In Ethiopia, the level of domestic violence against women is one of the highest in the world. However, Ethiopia is signatory for various conventions and incorporate into the constitution and other legal frameworks. Nevertheless, effective implementation of the existing policy documents, and engaging different stakeholders is very limited. There is paucity of evidence on piloting the feasibility of implementing community based preventive intervention programs. Therefore, the main aim of this study is to pilot feasibility and implement existing research evidence and policy documents at community level to prevent domestic violence against women in Awi zone, northwestern Ethiopia This study will be conducted in three districts of the Awi zone, Amhara regional state, Northwestern Ethiopia.

General Objective:The overall aim of this study is to assess the outcome of community based interventions implementation to prevent domestic violence against women, enhance community response and determinants among women (15-49 years) in Awi Zone, Northwestern Ethiopia from November, 2017 to November, 2018.

Specific Objectives

1. To assess the baseline level of domestic violence against women in the study area
2. To identify associated factors of domestic violence against women
3. To design intervention implementation strategy to tackle domestic violence against women
4. To implement culturally appropriate/acceptable interventions to address bottlenecks and domestic violence against women
5. To assess the outcome of community based intervention on domestic violence against women

Research questions

* How can prevent domestic violence against women through community based intervention?
* What are the bottlenecks of prevention intervention implementation at community level?
* How can implementers engage stakeholders to mobilize community and resource to implement existing evidence based interventions to transform gender norm?

Research Hypothesis

* Null hypothesis (Ho): this community based prevention intervention will not have effect (difference) on the level of domestic violence against women as compared with control (standard program).
* Alternative Hypothesis (HA): community based prevention intervention will have a better effect to make an improvement on the level of domestic violence against women than control (standard services).

DETAILED DESCRIPTION:
Sample Size Determination The sample size is determined considering both the intervention and control group proportion. The sample size for dichotomous outcome is recommended based on an assumption of superiority trial hypothesis testing. The hypothesis of the researcher is that implementation of the new community based prevention intervention program to prevent domestic violence against women will have significant effect than the standard (existing) prevention program in public health point of view. So the corresponding null hypothesis (Ho) is that: the new community based preventive intervention is not more efficacious to prevent domestic violence against women than the comparison group based on public health relevance. In addition, the sample size is determined considering an assumption of 5% margin of error, 95% significance level and 80% power.

Where; N is the sample size of each group, P is prevalence in standard intervention/control arm, d: the real difference between two treatment effect (d= Po-Px); 22%-9%=13%=0.13); δ0: a statistical acceptable margin (5%); ɑ: is the significance level which is 95% confidence level (ɑ=1-0.95=0.05=1.645), ß: is 80% power (ß=1-0.8= 0.2 = 0.845, and adding Then, considering 10% for potential non-achieved rate compensation. The calculated sample size for a group is 364. Eventually, as a result of the complex sampling design (multistage, stratified and systematic sampling), design effect is considered increase power and precision of the study. Design effect was computed using a finding from complex sampling design study conducted in Ethiopia (Fagitalekoma district) reported that the prevalence of DVAW was 78%, and a clustered randomized control trial done in Uganda indicated that 22% of women experienced physical IPV in the standard intervention group. The final sample size for the three arms was 1,758 women that mean 586 for each group. The number of participant in the qualitative study will be determined by information saturation during interviews and or focused group discussions (FGD). A minimum of two FGD (one male group and one female group) which comprise 8 to 10 discussants will be held at each selected kebeles. The local leaders or other person who are in-charge will be participated on the selection of qualitative study participants until information saturation.

Sampling Procedure

Multistage, stratified and systematic sampling will be used to select study participant to this study. First, contextual assessment will be employed among purposefully selected study participants from Awi zonal admisntration, district offices and community representatives. Stakeholders such as local politicians, health office, women and children affair office in-charges, local leaders, police, health care providers, non-governmental organization representatives and other concerned bodies will be participated to involve on advocacy meeting and contextualization. Then, multi-stage stratified probability sampling methods will be used to select study sites (kebeles) in the three districts among nine districts in Awi zone. Three districts will be selected for three experimental group. One district will be selected for comprehensive intervention. The second district will be assigned for partial intervention group, and the third district will be taken as comparison (control). Then, six kebeles (two kebeles from each district) will be selected from three districts purposefully considering appropriateness for intervention, resource, and geographical proximity to control information contamination between intervention and control group.

Then, kebeles will be stratified into urban and rural Kebele in respective district. Stratification will use to control the awareness level, access to information, and community tradition gender norm variability between urban and rural dwellers. After that, proportional to size allocation (ni) of the sample size will be done to each stratum. Eventually, systematic sampling will be employed to select actual study participants at household level based on kth interval. Confidential code will be given strictly to households that will be selected for interview for intervention monitoring and endline evaluation purpose. In the meantime, if two married women present in one household with one husband (polygamy), only one woman will be selected using lottery method for interview.

Regarding to qualitative study, purposive sampling method will be used to select study participants for in-depth interview, key informant interview (KII) and FGD. The community leaders will be consulted and actively involved on the recruitment of the most knowledgeable and respected community representatives for in-depth interview, key informant interview (KII) and FGD. The purpose of the study will be explained in detail to the community leaders who will participate on the recruitment of qualitative study participants. It will be conducted to assess individual perception towards DVAW mainly focused on sex negotiation, decision making, community gender norm, and wife beating attitudes with in the community. In addition, community sanction (response) against DVAW will be assessed qualitatively. It will mainly involve by taking from people who are in position (authority) such as local leaders, religious fathers, elders, police, women affair office, women association, health professionals, health extension workers, and women lawyers.

Data Collection

Mixed data collection method will be carried out using structured and semi structured questionnaires, that adapted from various literature. The tool will be pretested, modified to the local context and suite to the study objectives. The tool will consisted of demographic, socio-economic characteristics of couples (women self-reported profile), relationship level, community level and societal level factors of domestic violence. In addition, the tool will comprise questions about the experience of psychological, physical, sexual violence. In addition, semi structured questionnaire will be designed for qualitative study. Similarly, interview guide will be used to assess and dig-out the underlying bottlenecks in the community that hinder implementation of preventive interventions.

Data Collection Procedure

Data will be collected using sequential explanatory mixed method for baseline, intervention monitoring/tracking and endline implementation evaluation. Here below is the flow chart of the mixed data collection process adapted from other study. Two quantitative (1 and 2) and qualitative (1 and 2) process will be sequentially implemented to gather necessary data . Face-to-face interview method among married or cohabited women, key informant interview, in-depth interview, focus group discussion, meeting and training time data capturing will be carried out to have relevant information. In addition to the domestic violence assessment tool, the alternative questionnaire will be prepared and provide to data collectors to secure confidentiality issue if incase of third person might come suddenly during interview time. Very confidential place for women will be arranged by data collectors as per the training and WHO VAW research ethics recommendation.

Then qualitative data collection (KII, in-depth interview and FGDs) will be held to explore community perception, attitudes, norms and beliefs about domestic violence. However, mini (quick) qualitative data collection for contextualization has been done among officially in the districts and zone administrative level. On the other hand, it will use to find out community mobilization strategies, existing legal sanctions, available training guidelines, collaboration and integration of implementation activity. This will also help to design appropriate tool for main study, to design correct and culturally compatible intervention materials to tackle the problem. The KII will be held among women representative, district council members, women affair office, police officers, lawyers, elders, local politicians/leaders, health care providers, nongovernmental organization, and religious leaders.

Gender specific focused group discussion will be held on group of men and women to assess societal perception about domestic violence against women. Each focus group discussion will consisted of eight to ten participants. All participants' sociodemographic data will be captured using anonymously coded structured questionnaire. The FGDs will be facilitated by a group of three people (moderator, note taker and principal investigator). Voice recorder, note taking and nonverbal communication (physical gestures) during the discussion will be recorded as much as possible to capture necessary information. An estimate of 60 to 90 minutes will be taken to conduct one FGD. Moreover, implementation of domestic violence against women preventive intervention activities will be monitored/tracked using ongoing qualitative study method. Eventually, intervention implementation endline evaluation will be carried out using as same structured questionnaire, data collectors and supervisors as of the formative assessment. Data will be collected by exclusively twelve female health professionals (Nurse, Midwifery or public health).

Data Quality Assurance

Participants Allocation: Allocation of study participants in the intervention and control group will be considered geographic proximity to minimize information contamination. Representative sample will be taken using scientifically sounded procedures.

Appropriate Data Collectors recruitment: Data will be collected by twelve trained Diploma and above qualification female Nurses, Midwives and or public health officers who are not local resident in the community for trustworthiness and ethical concerns. Four supervisor who have Master of Public Health (MPH) with good previous field survey experience will be recruited.

Data Collectors Training: A five days training will be given for research assistants by the principal investigator. The training will mainly focus on the purpose of the study, data collection procedure, interview techniques, sampling methods, strict protection of confidentiality, ethical issues of VAW research and data quality assurance. Ethical sensitiveness of VAW will be explained to research assistants to maintain confidentiality and also quality of data. Brief explanation will be provided on biomedical research ethical principles and WHO (2001) gender based violence research ethical guideline recommendations called "women's safety first". Refreshment training and short orientation/debriefing will be provided regularly to research assistants during the study period.

Pretest: Pretest will be done among 5% of the sample size among married women from nearby district to check the compatibility of the data collection tool. The pretest will address sensitive words in the question, time, data collection procedure, interview techniques, sequence of questions, consent taking from study participants, and FGD facilitation skill and note taking. Necessary amendment will be taken according to feedback from study participant (verbal and non-verbal expression during pretest interview) and comment from research assistants.

Training of Implementers: intensive training and supportive supervision will be given for implementers. Two implementation facilitators and 6 community health extension workers will be recruited and hired for one year (12 months) contract employment. Implementers will be participated on the intervention tool validation to be familiar with the tool. Regular discussion and close supportive supervision will be given by principal investigator and facilitators.

Data Processing and Statistical Analysis

Baseline, monitoring and end-line gathered data will be checked and edited for incompleteness and inconsistency at field as well as at office. Explanatory and outcome variables will be clearly predefined prior to data entry. During data entry if woman will report at least one type of experience of either physical, psychological or sexual violence items coded as "Yes = 1" and "No = 0". On the other hand, women acceptance to violence or gender inequity norm will be measured using six questions/measurements, and also if women respond at least one justifies of wife beating. Similarly women autonomy will be measured in four components autonomy indicators such as women's economic decision-making autonomy, familial health care and family planning decision-making autonomy, extent of freedom of movement autonomy, and women's attitudes toward partner's violence. After completing the definition and coding of raw data. Data entry template will be designed on Epi data window version 3.5.1, and data entry will be carried out.

Then data will be exported to SPSS window version (23.0) for further analysis. Data cleaning will be performed computing frequency using box plot to explore outliers and other data anomalies. Multiple imputation will be done to handle missing data. Different statistical assumptions will be checked for data distribution and suitability for statistical analysis. Descriptive statistics will be computed to determine prevalence (proportion), mean, median, and standard deviation of some independent variables as necessary. Cross tabulation (chi-square) will be employed. Binary logistic regression will be carried out to confirm the association of explanatory variable with DVAW. Explanatory variable which will have score of p-value less than 0.25 in binary logistic regression will be included into the multiple logistic regression analysis to determine the independent determinants of domestic violence by controlling the confounding variable. In addition, Intention to Treat Analysis (ITTA) will be carried out to compute the overall changes on the level of DVAW. Moreover, Difference in Difference (DID) will be calculated to determine the net intervention effect. The DID will be computed as subtracting intervention arm outcomes from baseline data to endline minus difference of control arm outcomes from baseline to endline. Finally, statistical significance of intervention effect will be measured using adjusted prevalence ratio, adjusted odd ratio/adjusted risk ratio at 95% CI and p value less than 0.05.

Qualitative data will be transcribed through playing and replaying the voice recorder and also referring the note taken during interview or FGD. The voice recorder audio will be listen multiple times as much as possible at very quiet place. It will be transcribed independently by research assistant and principal investigator according to the verbatim of participants. Then transcribed qualitative data will be translated from local language (Amharic) into English. In the meantime, the qualitative data will be read and reread to understand what they want to say. The quotes will be narrated and cited using participant's code. All the qualitative data gathered from interview and FGD will be arranged into thematic areas. Similar ideas will be color coded, and then merged accordingly. Qualitative Data Analysis (QDA) software like Nvivo will be used to arrange or organize manually coded qualitative data.

ELIGIBILITY:
Inclusion Criteria

* Both the intervention and control participants will be selected from the general population
* All married and or cohabited women (15-49 year)
* Got married and stayed with partner at least 12 months
* Registered or recognized as permanent (at least 6 months)

Exclusion Criteria

- participants who are unable to respond due to severe physical or mental illness

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 1217 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the level of domesic violence against women from baseline to endline assessent | 12 month period from baseline assessment to endline interevntion evalaution
  The primary outcome is a change on domestic violence agaianst women. The main measure is the change in the prevalnce of domestic violence, engament of stakeholders, integration of the prevention intervention with existing community health program and the level of awarenss of the community about gender equality.

CONTACTS AND LOCATIONS:
Overall Officials: Augustine Ankomah, PhD, Study Chair — University of Ghana; Kwasi Torpey, MD, PhD, Study Chair — University of Ghana; Abubakar Manu, PhD, Study Chair — University of Ghana
Locations (1):
- Awi zone administaration, Injibara, Amhara Regional State, Ethiopia

REFERENCES:
- [Derived] Semahegn A, Torpey K, Manu A, Assefa N, Ankomah A. Community based intervention to prevent domestic violence against women in the reproductive age in Northwestern Ethiopia: a protocol for quasi-experimental study. Reprod Health. 2017 Nov 21;14(1):155. doi: 10.1186/s12978-017-0414-2. PMID 29162117